CLINICAL TRIAL: NCT05688527
Title: The Effects of a 5-Step Skin Regimen on Pigmentation and Appearance Related Biophysical Properties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Arbonne (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARB_SKIN5
Record Dates: First submitted 2023-01-05; First posted 2023-01-18 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5 Step Skin Care Regimen (Experimental): The subject uses 5 facial products in the regimen; a cleansing balm, a toner, a serum, a moisturizer and an eye cream.
  Interventions: Other: Cleansing Balm; Other: Toning Essence; Other: Facial Serum; Other: Moisturizer; Other: Eye Cream

INTERVENTIONS:
Other: Cleansing Balm — DermResults Cleansing Balm w/ Avocado Oil twice daily
Other: Toning Essence — DermResults Advanced Toning Essence w/ Mineral Booster twice daily
Other: Facial Serum — DermResults Advanced Serum w/ Hyaluronic Acid twice daily
Other: Moisturizer — DermResults Advanced Moisturizer w/ Hyaluronic Acid twice daily
Other: Eye Cream — DermResults Advanced Eye Cream w/ Hyaluronic Acid twice daily

SUMMARY:
This study is to analyze the effects of a 5-step skin care regimen on various skin parameters such as pigmentation, and firmness and elasticity of the skin around the eyes. The 5 facial products in the regimen are a cleansing balm, a toner, a serum, a moisturizer. and an eye cream.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 35 years old and 65 years old.
* Must have fine lines and wrinkles around the eyes.

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding.
* Prisoners
* Adults unable to consent
* Individuals who have changed any of their hormonal based contraception within 3 months prior to joining the study.
* Subjects using any topical retinoid, hydroquinone, kojic acid, bakuchiol, hyaluronic acid or benzoyl peroxide containing topical product within 2 weeks of starting study or any subject unwilling to refrain from washout prior to enrollment.
* Subjects with any facial treatments in the past 6 months and who are unwilling to withhold facial cosmetic treatments during the study including botulinum toxin, injectable fillers, microdermabrasion, intense pulsed light (IPL), peels, laser treatments, acid treatments, tightening treatments, facial plastic surgery, or any other medical treatment administered by a physician or skin care professional which is designed to improve the appearance of facial skin.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-12-16 (Estimated)

PRIMARY OUTCOMES:
Appearance of facial wrinkles | 8 weeks
  Change in wrinkle severity measured by photographic analysis (BTBP 3D Camera System)
Change in skin pigmentation in the undereye area | 8 weeks
  Change in skin pigmentation in the undereye area by Skin colorimetric analysis of pigment

SECONDARY OUTCOMES:
Skin hydration | 1 week
  Change in skin hydration by SkinMoistureMeterSC measurement
Skin hydration | 4 weeks
  Change in skin hydration by SkinMoistureMeterSC measurement
Skin hydration | 8 weeks
  Change in skin hydration by SkinMoistureMeterSC measurement
Transepidermal water loss | 1 week
  Change in transepidermal water loss measurement with Vapometer
Transepidermal water loss | 4 weeks
  Change in transepidermal water loss measurement with Vapometer
Transepidermal water loss | 8 weeks
  Change in transepidermal water loss measurement with Vapometer
Skin volume | 1 week
  Change in skin volume/plumpness by photographic image analysis with BTBP 3D Camera System
Skin volume | 4 weeks
  Change in skin volume/plumpness by photographic image analysis with BTBP 3D Camera System
Skin volume | 8 weeks
  Change in skin volume/plumpness by photographic image analysis with BTBP 3D Camera System
Skin texture/roughness | 1 week
  Change in the appearance of photographic analysis of texture/roughness with BTBP 3D Camera System
Skin texture/roughness | 4 weeks
  Change in the appearance of photographic analysis of texture/roughness with BTBP 3D Camera System
Skin texture/roughness | 8 weeks
  Change in the appearance of photographic analysis of texture/roughness with BTBP 3D Camera System
Self-perception of skin parameters | 1 week
  Survey based self-assessment of facial fine lines and wrinkles, skin smoothness, skin firmness
Self-perception of skin parameters | 4 weeks
  Survey based self-assessment of facial fine lines and wrinkles, skin smoothness, skin firmness
Self-perception of skin parameters | 8 weeks
  Survey based self-assessment of facial fine lines and wrinkles, skin smoothness, skin firmness
Tolerability of products | 1 week
  Questionnaire based self-assessment about the tolerability of the topical skin products
Tolerability of products | 4 weeks
  Questionnaire based self-assessment about the tolerability of the topical skin products
Tolerability of products | 8 weeks
  Questionnaire based self-assessment about the tolerability of the topical skin products
Appearance of facial wrinkles | Change in wrinkle severity measured by photographic analysis (BTBP 3D Camera System)
  4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No